CLINICAL TRIAL: NCT06285903
Title: Comparing the Hydrodynamic Piezoelectric Technique With Osseodensification for the Assessment of Internal Sinus Iift-ing: (a Randomized Clinical Trial)
Brief Title: Comparing the Hydrodynamic Piezoelectric Technique With Osseodensification for the Assessment of Internal Sinus Iift-ing
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Shaymaa Hussein Rafat Kotb, Assistant lecturere of oral medicine ,periodontology departement at sphinx university, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUAREC20220002-11
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Bone Density, Low
Keywords: Dental implant; Osseointegration; primary implant stability; , internal sinus lifting; osseodensification,; piezoelectric
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: A total of 20 patients were randomly divided into two groups: Group1: patients received dental implant using osseodensification via Densah bur, Group2: patients received dental implant using hydrodynamic piezoelectric sinus lifting. The patients in both groups underwent bone grafting under sinus membrane. Modified bleeding index and probing depth were evaluated at 3, 6 and 12months intervals. An Osstell device was used to de-termine implant stability by recording the values of implant stability quotient (ISQ) im-mediately after implant placement and after 3 months. CBCT was performed before, af-ter 6 months and after 12 months to evaluate ridge height, bone density. Marginal bone loss was evaluated after 3 months via periapical radiograph, after 6 months and after 12 months via CBCT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Densah Bur (Experimental): patients received dental implant using osseodensification via Densah bur
  Interventions: Procedure: internal sinus lift surgery
- Group piezoelectric (Experimental): patients received dental implant using hydrodynamic piezoelectric sinus lifting
  Interventions: Procedure: internal sinus lift surgery

INTERVENTIONS:
Procedure: internal sinus lift surgery — surgery approach

SUMMARY:
Successful osseointegration considered the cornerstone in implant stability which predict the highest implants success outcomes. Implant stability depend on many factors like the implant design, surgical technique, and bone density. Posterior maxilla considered as a challenging area in implant placement, this is due to less dense trabecular bone sur-rounded by a thin layer of cortical bone which result in suffering in implant stability. The aim of this study is to evaluate the bone density outcomes using bone densification technique and piezoelectric surgical technique in sinus lift to promote bone gain

DETAILED DESCRIPTION:
Objectives: This study was directed to compare the outcomes of internal sinus lifting between osseodensification approach and piezoelectric surgery approach on the primary stability and osseointegration of dental implant.

Background data: Successful osseointegration considered the cornerstone in implant sta-bility which predict the highest implants success outcomes. Implant stability depend on many factors like the implant design, surgical technique, and bone density. Posterior maxilla considered as a challenging area in implant placement, this is due to less dense trabecular bone surrounded by a thin layer of cortical bone which result in suffering in implant stability. The aim of this study is to evaluate the bone density outcomes using bone densification technique and piezoelectric surgical technique in sinus lift to promote bone gain.

Materials and Methods: A total of 20 patients were randomly divided into two groups: Group1: patients received dental implant using osseodensification via Densah bur, Group2: patients received dental implant using hydrodynamic piezoelectric sinus lifting. The patients in both groups underwent bone grafting under sinus membrane. Modified bleeding index and probing depth were evaluated at 3, 6 and 12months intervals. An Osstell device was used to determine implant stability by recording the values of implant stability quotient (ISQ) immediately after implant placement and after 3 months. CBCT was performed before, after 6 months and after 12 months to evaluate ridge height, bone density. Marginal bone loss was evaluated after 3 months via periapical radiograph, after 6 , 12 months via CBCT.

ELIGIBILITY:
Inclusion Criteria:

free of systemic disease bone height at the site of the implant is ≤ 6 mm. have good oral hygiene.

-

Exclusion Criteria:

systemic diseases active periodontal disease , limited mouth-opening ability maxillary sinus disease or previous sinus surgery were also excluded smokers pregnant

Ages: 35 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Implant stability using the Osstell device by percentage | baseline ,3 months
  Primary implant stability (ISQ)

SECONDARY OUTCOMES:
Modified sulcus bleeding index,Peri-implant pocket depth (PPD)by mm | 3,6,9 months
  Clinical evaluation

OTHER OUTCOMES:
Bone Densityby mm | 3,6,12 months
  Crestal Bone Loss (CBL)

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Hammad Ibrahim, lecturer, Study Director — Al-Azhar University; Khalid s Hassan, Dean of Badr University, Study Chair — Faculty of Dentistry ,Badr university ,Assuit branch ,Egypt
Locations (1):
- Alazhar university ,Assuit branch ,Egypt, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Comparing the Hydrodynamic Piezoelectric Technique with Osseodensification for the Assessment of Internal Sinus Iift-ing: (a Randomized Clinical Trial)
Supporting Information: SAP
Time Frame: 1 month
Access Criteria: DOI:10.21203/rs.3.rs-4132878/v1
URL: https://papers.ssrn.com/sol3/papers.cfm?abstract_id=4759103

REFERENCES:
- See also: orchid — https://orcid.org/my-orcid?orcid=0000-0002-8404-438X
- See also: researchgate — https://www.researchgate.net/profile/Shimaa-Hussein-Kotb
- See also: web of science — https://www.webofscience.com/wos/author/record/ABE-1539-2022